CLINICAL TRIAL: NCT06567808
Title: Prevention of Infections in Cardiac Surgery (PICS): a Cluster-randomized Factorial Cross-over Trial
Acronym: PICS
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: PICS
Record Dates: First submitted 2024-08-20; First posted 2024-08-23 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2024-08

CONDITIONS: Infection, Surgical Site
MeSH Terms: conditions — Surgical Wound Infection | interventions — Cefazolin; Vancomycin

STUDY DESIGN:
Intervention Model Description: Factorial Assignment
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- cefazolin short-term (Experimental): Cefazolin 2g (or 3g if greater than 120kg body weight) will be given within an hour of surgery. The intraoperative dose at 4 hours after the first dose or upon wound closure (whatever comes first).
  Interventions: Drug: Cefazolin
- cefazolin long-term (Experimental): Cefazolin 2g (or 3g if greater than 120kg body weight) will be given within an hour of surgery. The intraoperative dose at 4 hours after the first dose or upon wound closure (whatever comes first) and the five post-operative doses in the long-term arms will be 2g every 8 hours.
  Interventions: Drug: Cefazolin
- cefazolin plus vancomycin short-term (Experimental): Cefazolin 2g (or 3g if greater than 120kg body weight) will be given within an hour of surgery. The intraoperative dose at 4 hours after the first dose or upon wound closure (whatever comes first). Vancomycin will be dosed at roughly 15mg/kg body weight intravenously, i.e. 1g or 1.5g if greater than 85kg body weight and is to be administered within 60-90 minutes of the surgical procedure.
  Interventions: Drug: Cefazolin; Drug: Vancomycin
- cefazolin plus vancomycin long-term (Experimental): Cefazolin 2g (or 3g if greater than 120kg body weight) will be given within an hour of surgery. The intraoperative dose at 4 hours after the first dose or upon wound closure (whatever comes first) and the five post-operative doses in the long-term arms will be 2g every 8 hours. Vancomycin will be dosed at roughly 15mg/kg body weight intravenously, i.e. 1g or 1.5g if greater than 85kg body weight and is to be administered within 60-90 minutes of the surgical procedure. The same dose will be used for the 3 post-operative doses in the long-term arm.
  Interventions: Drug: Cefazolin; Drug: Vancomycin

INTERVENTIONS:
Drug: Cefazolin — administration as outlined
  Other Names: Kefzol; Ancef
Drug: Vancomycin — administered as outlined
  Other Names: Vancocin; Firvanq
  Arms: cefazolin plus vancomycin long-term; cefazolin plus vancomycin short-term

SUMMARY:
The goal of this pragmatic, multi-centre factorial cluster randomized cross-over trial is to assess the efficacy of a combination of cefazolin plus vancomycin compared to cefazolin monotherapy, as well as a comparison of short versus long-term prophylaxis with four study arms: 1) cefazolin short-term, 2) cefazolin long-term, 3) cefazolin plus vancomycin short-term and 4) cefazolin plus vancomycin long-term.

DETAILED DESCRIPTION:
Although antibiotic prophylaxis is considered the cornerstone of prevention for sternal surgical site infections (s-SSIs), the most effective antimicrobial regimen and optimal duration remain unclear. There is a pressing need to determine how best to prevent sternal surgical site infections and at the same time reduce adverse events from unnecessary antibiotic exposure. Currently, due to the lack of evidence, unproven approaches prevail and adherence to guidelines is poor. Rigorous randomized controlled trials data are needed for improved patient care.

A factorial cluster randomized cross-over trial, a design not used previously in this field, will address these gaps. To date, we have successfully enrolled close to 6,000 eligible patients in the vanguard study, and have shown that the trial as planned is feasible and operationally highly cost-effective.

ELIGIBILITY:
Inclusion Criteria:

Adult patients (≥18 years of age) undergoing open-heart surgery (i.e. sternotomy, including minimally-invasive surgical techniques through mini-sternotomies)

Exclusion Criteria:

1. On systemic antibiotics or with an active bacterial infection at the time of surgery
2. Previously enrolled in this trial
3. Known to be colonized with methicillin-resistant staphylococcus aureus (MRSA). Where it is unethical to not administer glycopeptides.
4. Beta-lactam or vancomycin allergy precluding the use of cefazolin or vancomycin, respectively
5. Participation in other studies that may interfere with this trial.
6. Patients undergoing cardiac transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 38000 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2028-04-30 (Estimated); Study Completion 2028-07-30 (Estimated)

PRIMARY OUTCOMES:
Deep incisional or organ/space (complex) sternal surgical site infection (CDC/NHSN) | 3 months post-surgery
  Sternal surgical site infections are defined by clinical and microbiological criteria of infection at the surgical site that are associated with the operative procedure occurring within 90 days after surgery.

SECONDARY OUTCOMES:
All types of sternal surgical site infections (superficial, deep, organ; (CDC/NHSN) | 3 months post-surgery
  Sternal surgical site infections are defined by clinical and microbiological criteria of infection at the surgical site that are associated with the operative procedure occurring within 90 days after surgery.
Clostridium difficile infection | 3 months post-surgery
  Laboratory confirmed
Mortality | 3 months post-surgery
  Mortality in participants with an active infection
Number of patients with acute kidney injury | 7 days post surgery
  Acute kidney injury following the Acute Kidney Injury Network definition
Number of patients with sternal revision surgery | 3 months post surgery
  For suspected sternal surgical site infection
Rate of antimicrobial resistant organisms causing sternal wound infections | 3 months post-surgery
  including relevant susceptibilities and stratified by study arm

CONTACTS AND LOCATIONS:
Overall Officials: Dominik Mertz, MD, MSc, Principal Investigator — Hamilton Health Sciences Corporation